CLINICAL TRIAL: NCT02421276
Title: Depressed AIRE Gene Expression Causes Immune Cell Dysfunction & Autoimmunity in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-2300
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Down Syndrome; Polyendocrinopathies, Autoimmune; Respiratory Tract Infections; Autoimmunity
MeSH Terms: conditions — Down Syndrome; Polyendocrinopathies, Autoimmune; Respiratory Tract Infections; Autoimmune Diseases | interventions — Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persons without Down syndrome (Other): White blood cell analysis from persons without Down syndrome assessed by absence of trisomy 21.
  Interventions: Other: Phlebotomy
- Persons with Down syndrome (Other): White blood cell analysis from persons with Down syndrome assessed by presence of trisomy 21.
  Interventions: Other: Phlebotomy

INTERVENTIONS:
Other: Phlebotomy — White blood cell analysis: Subtypes of white blood cells will be counted by flow cytometry

SUMMARY:
This study plans to learn more about Down syndrome. The investigators think there is a different level of the AIRE gene in individuals with Down syndrome. The investigators think that the AIRE gene level can provide more insight about depressed immune cell function in individuals with Down syndrome. Patients are being asked to be in this research study because the investigators want to see if their blood contains more of less of the AIRE gene.

DETAILED DESCRIPTION:
Down Syndrome (DS) is the most common chromosomal abnormality among live-born infants. Through full or partial trisomy of chromosome 21, DS is associated with cognitive impairment, congenital malformations (particularly cardiovascular), and dysmorphic features. In addition, immunological abnormalities are much more prevalent in individuals with DS. For example, DS is associated with increased susceptibility to infection, as revealed in 2009 during the influenza pandemic where the likelihood of death was 300 times greater for DS patients than the general population. DS patients have increased frequencies of autoimmune disorders and leukemias, yet curiously, have a decreased risk for allergic diseases, particularly asthma. Perhaps the most telling statistic for immunologic abnormality in DS patients is that respiratory tract infections are the most important cause of mortality in DS at all ages.Our studies have identified AIRE as a master control gene that is aberrantly decreased in persons with DS, leading to autoimmunity and immunologic abnormalities. AIRE ("autoimmune regulator"), although encoded on chromosome 21, is also significantly reduced in expression in DS, where it may contribute to autoimmune and immune dysregulation. The investigators will test the hypothesis that immune dysfunction and autoimmune disease preferentially occur in DS as a consequence of deficient expression of AIRE in peripheral blood cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age newborn up until the twenty-second birthday.
2. Diagnosed with idiopathic or secondary pulmonary arterial hypertension as defined by a mean pulmonary artery pressure > 25 mmHg at rest or > 30 mmHg with exercise.
3. Confirmed trisomy 21.
4. Followed by the Pulmonary Hypertension Program and Sie Center at The Children's Hospital.
5. The investigator or co-investigator must obtain written informed consent and assent where applicable before any study procedure is performed or data is collected.

Exclusion Criteria:

1. Any person older than 22 years of age
2. Patients with sickle cell disease with Pulmonary Arterial Hypertension (PAH) as treatment is defined differently within this population.
3. In the opinion of the investigator, a patient who is unlikely to cooperate or complete the study for any reason.

Max Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
AIRE Gene expression in Macrophage Subpopulations | At the time of sample acquisition
  Peripheral blood draw

SECONDARY OUTCOMES:
White blood cell Subpopulation Numbers | At the time of sample acquisition
  Peripheral blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Yeager, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Denver, Denver, Colorado, United States